CLINICAL TRIAL: NCT05058274
Title: Clinical Results of a Monofocal Aspheric Bitoric Intraocular Lens With Plate Haptics in Hyperopic Eyes (HIPER-AT-TORBI)
Acronym: HIPER-AT-TORBI
Status: Completed | Type: Observational
Sponsor: OFTALVIST (Oftalmología Vistahermosa S.L) (Industry)
Collaborators: Carl Zeiss Meditec AG (Industry)
Responsible Party: Sponsor
Other Study IDs: HIPER-AT-TORBI
Record Dates: First submitted 2021-09-08; First posted 2021-09-27 (Actual); Last update posted 2024-03-22 (Actual); Status verified 2024-03

CONDITIONS: Astigmatism; Far Sightedness; Cataracts
MeSH Terms: conditions — Astigmatism; Hyperopia; Cataract

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No

GROUPS / COHORTS (1):
- Single arm: All participants
  Interventions: Device: Implant of the AT-TORBI 709 lens

INTERVENTIONS:
Device: Implant of the AT-TORBI 709 lens — Implant of the AT-TORBI 709 lens

SUMMARY:
Observational post-marketing study with prospective follow-up of CE marked medical devices aimed at the treatment of hyperopia and astigmatism in patients with cataract. The objective is to evaluate the clinical results of the implantation of the monofocal aspheric bitoric intraocular lens (IOL) with AT-TORBI 709 plate haptics in cataract surgery of hyperopic eyes with astigmatism.

DETAILED DESCRIPTION:
All patients participating in the study will have the intraocular lens (IOL) AT TORBI 709 implanted from Carl Zeiss Meditec AG, Jena, Germany, with CE marking. All patients will be treated according to standard clinical practice. A preoperative and postoperative evaluation will be carried out one month, six and twelve months after the intervention where the following tests will be performed: refraction, corneal topography, measurement of visual acuity with and without correction, slit lamp examination, eye biometry using the IOLMaster 700 Carl Zeiss Meditec AG, Jena, Germany, CE marked optical non-contact biometer, contrast sensitivity with the CC-100 screen (Topcon Europe, The Netherlands), and the Catquest-9SF (European Registry of Quality Outcomes for Cataract and Refractive Surgery, founded by the European Society of Cataract and Refractive Surgeons). The sponsor has received an unrestricted research grant by Zeiss.

ELIGIBILITY:
Inclusion Criteria:

1. Patients of 50 years of age or older to undergo cataract surgery with phacoemulsification
2. Patient who signs the informed consent.
3. Regular corneal astigmatism between 1.0D and 4.0D.
4. IOL power between 21D and 26D
5. Target-target distance measured with the IOLMaster 700 biometer (Carl Zeiss Meditec AG) greater than 11.6 mm.
6. Patients with hyperopia between 1.0D and 4.0D.

Exclusion Criteria:

1. Patients who do not provide informed consent
2. Patients who do not understand the study procedure
3. Previous corneal surgery.
4. Irregular cornea (eg keratoconus)
5. myopic patients
6. Eye abnormalities or pathologies that could reduce the visual function or stability of the IOL (eg severe amblyopia or macular degeneration)

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who are going to undergo conventional cataract surgery by phacoemulsification following regular clinical practice and present hyperopia with astigmatism.
Sampling Method: Non-Probability Sample
Enrollment: 60 (Actual)
Dates: Start 2021-11-03 (Actual); Primary Completion 2024-02-21 (Actual); Study Completion 2024-02-21 (Actual)

PRIMARY OUTCOMES:
Measurement of the refractive error | 12 months
  Measurement of the refractive error (equivalent spherical error, the refractive cylinder and the astigmatism vectors (J0 and J45) )
Measurement of the rotational stability | 12 months
  Measurement of the rotational stability

SECONDARY OUTCOMES:
Measure of visual acuity | 12 months
  Measurement of visual acuity
Measure of corneal topography | 12 months
  Measure of corneal topography
Measure of ocular biometry | 12 months
  Measure of ocular biometry
Measure of contrast sensitivity | 12 months
  Measure of contrast sensitivity
Satisfaction questionaire | 12 months
  For several questions percentage of respondants answering each of five possible provided answers ranging progressively from strong disatisfaction to strong satisfaction (1-4) as well as an answer for those patients who cannot decide (5)
Slit lamp examination | 12 months
  Slit lamp examination

CONTACTS AND LOCATIONS:
Overall Officials: Pedro Tañá Rivero, Doctor, Principal Investigator — OFTALVIST (Oftalmología Vistahermosa S.L)
Locations (2):
- Spain (2):
  - OFTALVIST (Oftalmología Vistahermosa S.L.), Alicante
  - OFTALVIST (Oftalmología Vistahermosa S.L.), Valencia

IPD SHARING:
Plan to Share IPD: Undecided
A publication summarizing the results of the study will be made public after the study termination.